CLINICAL TRIAL: NCT03545373
Title: Randomised Controlled Clinical Trial Investigating Benefits of Using Response to Broad Spectrum Antibiotics as an Exclusion Diagnostic for Tuberculosis (TB) in Primary Care Adult Patients Versus Risk of Antimicrobial Resistance (AMR)
Brief Title: Accuracy and Consequences of Using Trial-of-antibiotics for TB Diagnosis (ACT-TB Study)
Acronym: ACT-TB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15232
Record Dates: First submitted 2018-05-01; First posted 2018-06-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Tuberculosis; Respiratory Tract Infections; Pneumonia
Keywords: antimicrobial resistance; TB; Cough; antibiotics; anti-infective agents
MeSH Terms: conditions — Tuberculosis; Respiratory Tract Infections; Pneumonia; Cough | interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Three treatment arms allocated using computer generated block randomization in a 1:1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: All laboratory forms for mycobacteriology and nasopharyngeal pneumococcal work will have no reference to participant treatment allocation. On Day-8, assessment of improvement from baseline symptoms will utilize audio computer-assisted self-interview (ACASI) to minimise potential for social-mediated reporting and ascertainment biases. On Day-29, clinical outcome assessment forms will bear no reference to treatment arm. Participants, research coordinators, and routine care staff will not be masked to ensure safety of the participants and allow appropriate patient management decision-making which may be related to the trial interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azithromycin (Experimental): Azithromycin 500mg, oral, once daily for 3 days commencing on randomization day.
  Interventions: Drug: Azithromycin
- Amoxicillin (Experimental): Amoxicillin 1g, oral, 3 times daily for 5 days commencing on randomization day.
  Interventions: Drug: Amoxicillin
- Standard of care (No Intervention): The standard of care in current national guidelines for patients presenting with cough and without danger signs (No treatment, re-evaluate with sputum results)

INTERVENTIONS:
Drug: Azithromycin — Azithromycin tablet taken orally
  Arms: Azithromycin
Drug: Amoxicillin — Amoxicillin tablets taken orally
  Arms: Amoxicillin

SUMMARY:
This is a three-arm, open-label individually randomised controlled clinical trial investigating the benefits of the diagnostic use of broad-spectrum antimicrobials during the diagnostic process for tuberculosis (TB) and the risk of antimicrobial resistance. Adults (≥18 years) presenting to primary care with TB symptoms will, after excluding acute illness, be randomised (1:1:1) to receiving azithromycin, amoxicillin or standard care. Diagnostic accuracy will be ascertained by comparing self-reported response to treatment on Day-8 to results of mycobacteriology tests (MTB culture, smear microscopy and Xpert/MTB/RIF). Antimicrobial resistance will be ascertained by comparing arms with respect to incidence of resistant Streptococcus pneumonia carriage cultured from nasopharyngeal swabs collected on Day-28. Clinical benefit will be ascertained by comparing clinical outcomes by Day-29.

DETAILED DESCRIPTION:
BACKGROUND

Antimicrobial resistance (AMR) is a growing public health threat that is in part fuelled by empirical antibiotic usage. Empirical antibiotic use is often motivated by lack of point of care diagnostics a common problem in infectious diseases most of which are life-threatening. Tuberculosis (TB), the leading cause of infectious disease mortality, is one of the life-threatening illnesses without adequate diagnostics. Just over 50% of TB cases reported to WHO annually have confirmed mycobacteriological diagnosis. To complement the diagnostic gap, standard diagnostic algorithms include empirical antibiotic use. The antibiotic course, referred to as "trial-of-antibiotics", given to mycobacteriology-negative but symptomatic adults, is often broad-spectrum aiming to provide treatment for pneumonia. The goal is to treat infectious causes of respiratory symptoms other than TB, effectively performing the role of a "rule-out" diagnostic test for TB.

RATIONALE

Approximately 26.5 million antibiotics courses are prescribed in the course of diagnosis of the 5.3 million smear negative TB registrations per annum. Despite this widespread use, there is no randomised controlled trial (RCT) evidence supporting the diagnostic accuracy of antibiotic trials and their impact on AMR. It is also unknown whether this usage of antibiotics can improve clinical outcomes considering that in settings of high HIV prevalence, bacterial infection associated mortality just before and during TB treatment is high.

OBJECTIVES

Primary

1. To establish the diagnostic value of trial-of-antibiotics for excluding pulmonary tuberculosis (PTB) in adults with prolonged cough (and have a valid sputum test result) at primary care level in Malawi.
2. To determine the overall clinical benefit of giving empirical antibiotic treatment in primary care participants with chronic cough.

   Secondary
3. To evaluate using nasopharyngeal Streptococcus pneumonia carriage, the effect of a trial-of-antibiotics on selection for antimicrobial resistance.
4. To establish the diagnostic value of trial-of-antibiotics for excluding pulmonary tuberculosis (PTB) in primary care presenting Malawian adults with prolonged cough including those without a successful sputum
5. To estimate the incremental cost-effectiveness of trial-of-antibiotics using azithromycin and trial-of-antibiotics using amoxicillin in comparison to standard of care, and to each other.

METHODS To address the evidence gaps related to a) accuracy, b) antimicrobial resistance, and c) impact on clinical outcomes), a randomised controlled clinical trial recruiting adult patients (≥18 years) presenting to primary care centres in Blantyre, Malawi with history of cough for at least 2 weeks, will be conducted. After excluding those with danger signs participants will be randomised to receiving or not receiving trial-of-antibiotics (azithromycin or amoxicillin) from Day-1 to determine diagnostic accuracy (specificity) against mycobacteriology reference standard (smear microscopy, Xpert/MTB/RIF and culture).

Differences in antimicrobial resistance and clinical outcomes [1)death, 2)hospitalisation, 3)missed TB diagnosis] will be compared between treatment arms by Day-29.

To adequately address these objectives, 388 sputum-TB-negative participants will be required for each of the three arms (azithromycin, amoxicillin and standard of care).

FUNDING

Funding was provided by Commonwealth Scholarship Commission (Titus Divala), Helse Nord RHF (Titus Divala), Wellcome Trust Senior Research Fellowship in Clinical Science (WT200901, Liz Corbett), and the UK Medical Research Council (MRC) and the UK Department for International Development (DFID) (MR/K012126/1, Katherine Fielding).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory clinic attendees presenting with cough
* Unwell for at least 14 days
* Aged at least 18 years
* Reside in Blantyre and willing to return to the same clinic for follow up visits over the entire study period.

Exclusion Criteria:

* Self-reported allergy to study medications
* WHO/Malawi National tuberculosis Program (NTP) danger signs: respiratory rate > 30/min, temperature >39oC, Heart rate >120/minute, confused/agitated, respiratory distress, systolic blood pressure <90 mmHg, inability to walk unassisted
* Treated with antibiotics other than co-trimoxazole prophylaxis within the past 14 days
* Tuberculosis treatment or isoniazid preventive therapy within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1583 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of trial-of-antibiotics: proportion of patients without tuberculosis (by sputum tests) who report improvement of their baseline illness when asked 7 days after randomisation (Day 8 study visit). | Day 1 to Day 8
  The proportion of patients without tuberculosis (by sputum tests) who report improvement of their baseline illness when asked 7 days after randomisation (Day 8 study visit).
  This can be thought of as diagnostic specificity if you take sputum test results as a reference standard and change in symptoms at Day 8 as the investigational test.
  In this case the possible results of the investigational test are improvement and no improvemet (no change or worsened) in response to the question: on day 1, you reported that you were unwell; compared to that day, has your illness worsened, remained the same, or improved?
  The mycobacteriology reference standard will be defined in participants with at least one valid sputum test result on days 1 and 8 as sputum-test-positive if there is at least one positive of smear microscopy, Xpert/MTB/RIF, or MTB culture; and as sputum-test-negative if none of the tests is positive.
Clinical impact of trial-of-antibiotics | Day 1 to Day 29
  We will investigate the overall clinical impact of trial-of-antibiotics by comparing the day 29 risk of any of
  1. death,
  2. hospitalisation, and
  3. missed tuberculosis
  The connection between trial-of-antibiotics and risk of hospitalisation and death assumes a protective effect of antibiotics. In patients presenting with chronic cough at primary care in high HIV prevalence settings, frequencies of mortality and hospitalization over a two months period are similar, ranging from 2 to 6%.
  We have included missed tuberculosis diagnosis because this too can lead to death. We are defining "missed tuberculosis" as participants who meet standard mycobacteriological and radiological tuberculosis definitions but are incorrectly classified as tuberculosis-negative and not yet on tuberculosis treatment by Day 29.

SECONDARY OUTCOMES:
Impact of trial-of-antibiotics on antimicrobial resistance | Day 1 to Day 29
  We will use Streptococcus pneumoniae isolated from swabs of the nasopharynx as the indicator pathogen for AMR evaluation. An ecological niche for many bacterial species, the upper respiratory tract also presents a convenient window for investigating antimicrobial resistance.
  We will define AMR positive as having nasopharyngeal isolates of Streptococcus pneumoniae that are resistant to any of the following commonly used antibiotics: ceftriaxone, amoxycillin, cefoxitin, azithromycin, and erythromycin as determined using disc diffusion technique; and AMR negative as either (1) not isolating any Streptococcus pneumoniae or (2) isolating any Streptococcus pneumoniae that is not resistant to any of the assessed antibiotics. For each arm, and at both baseline and day 29, we will report proportion of AMR positive participants. The study outcome will be the proportion of AMR positive participants at day 29.
diagnostic value of trial-of-antibiotics in all patients including those without a valid sputum result | Day 1 to Day 8
  In this analysis, all will remain as described for primary outcome 1 except for the denominator, which will now include those without a valid sputum test result. The mycobacteriology reference standard for secondary outcome 2 will be defined as sputum test positive if at least one positive of smear microscopy, Xpert/MTB/RIF, or MTB culture from samples collected on days 1 and 8.
  The reference test will be sputum-test-negative if none of the tests is positive and where there is no valid sputum test result available. The most likely reason for not having a valid sputum result will be inability to produce sputum, but other explanations will be: lost sample before laboratory analysis, an invalid laboratory reading, or contamination. We have opted to analyse this population because in symptomatic adults of the study setting, failure to produce sputum can be as high as 13%.
Economic analysis of use of trial-of-antibiotics | Day 1 to Day 29
  To estimate the incremental cost-effectiveness of trial-of-antibiotics using azithromycin and trial-of-antibiotics using amoxicillin in comparison to standard of care, and to each other using a combination of information from the following data:
  1. Incremental cost per quality adjusted life year gained
  2. Total direct medical costs per participant
  3. Eq-5D utility score

CONTACTS AND LOCATIONS:
Overall Officials: Titus H Divala, MBBS MPH MS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- University of Malawi College of Medicine, Blantyre, Southern Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Data sharing of all data with any group requesting access to individual records will be ensured within 12 months of completion of publication related analyses, with all data and study tools made available by that time through the institutional research data repository established by London School of Hygiene & Tropical Medicine(LSHTM) Research Data Management Support Service..
  Anonymised data will be held for sharing as original databases stored with a soft copy of the fully annotated questionnaires and the STATA files used for recoding and analysis. Personal identifiers, such as names, will not be held, with ID numbers used instead.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publishing study main papers.
Access Criteria: Through the London School of Hygiene & Tropical Medicine data repository.

REFERENCES:
- [Derived] Divala TH, Corbett EL, Kandulu C, Moyo B, MacPherson P, Nliwasa M, French N, Sloan DJ, Chiume L, Ndaferankhande MJ, Chilanga S, Majiga ST, Odland JO, Fielding KL. Trial-of-antibiotics to assist tuberculosis diagnosis in symptomatic adults in Malawi (ACT-TB study): a randomised controlled trial. Lancet Glob Health. 2023 Apr;11(4):e556-e565. doi: 10.1016/S2214-109X(23)00052-9. PMID 36925176
- [Derived] Divala TH, Fielding KL, Sloan DJ, French N, Nliwasa M, MacPherson P, Kandulu CC, Chiume L, Chilanga S, Ndaferankhande MJ, Corbett EL. Accuracy and consequences of using trial-of-antibiotics for TB diagnosis (ACT-TB study): protocol for a randomised controlled clinical trial. BMJ Open. 2020 Mar 25;10(3):e033999. doi: 10.1136/bmjopen-2019-033999. PMID 32217561